CLINICAL TRIAL: NCT05326828
Title: Implantable Cardiac Monitor to Detect Atrial Fibrillation in Patients With MINOCA
Acronym: MINOCA
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Zürich (Other); Bangerter-Rhyner Stiftung (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-D0009
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: MINOCA; Atrial Fibrillation
Keywords: Implantable cardiac monitor
MeSH Terms: conditions — MINOCA; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- ICM group: Patients eligible for ICM implantation for screening of atrial fibrillation
  Interventions: Device: CONFIRM Rx implantable cardiac rhythm monitor (Abbott); Diagnostic Test: Systematic etiologic work-up for underlying causes of MINOCA
- Non-ICM group: Patients ineligible for ICM implantation due to 1) refusal, 2) contraindication, or 3) clear underlying cause of MINOCA before ICM implantation.
  Interventions: Diagnostic Test: Systematic etiologic work-up for underlying causes of MINOCA

INTERVENTIONS:
Device: CONFIRM Rx implantable cardiac rhythm monitor (Abbott) — Implantation of CONFIRM Rx ICM
  Groups: ICM group
Diagnostic Test: Systematic etiologic work-up for underlying causes of MINOCA — Intracoronary optical coherence tomography, cardiac magnetic resonance imaging, transesophageal echocardiography, vasospasm testing, thrombophilia screening, Holter ECG (only non-ICM group)

SUMMARY:
Myocardial infarction with non-obstructive coronary arteries (MINOCA) (i.e.<50% stenoses) on coronary angiography) is an underappreciated clinical entity concerning 5-6% of patients with acute myocardial infarction. Approximately 50% of these patients remain without appropriate diagnosis and treatment.

The MINOCA study aims at systematically assessing the frequency of underlying pathologies of MINOCA and outcomes with a multidisciplinary etiologic work-up and follow-up of 5 years including, for the first time, an implantable cardiac monitor (ICM) to assess the frequency of atrial fibrillation as underlying cause for MINOCA.

DETAILED DESCRIPTION:
Approximately 5-6% of patients with acute myocardial infarction (AMI) have myocardial infarction with non-obstructive coronary arteries (MINOCA) (i.e.<50% stenoses) on coronary angiography and up to 50% of these patients remain without appropriate diagnosis and treatment. A multidisciplinary etiologic work-up of MINOCA has recently been proposed by international consensus documents. The present study aims for a structured scientific data collection from a full guideline-based work-up after MINOCA and follow-up of 5 years to assess clinical outcomes.

Untreated atrial fibrillation is a potentially neglected underlying cause of MINOCA. As implantable cardiac monitors (ICM) can detect atrial fibrillation with high accuracy, the aim of this study is, for the first time, to assess the occurrence of first diagnosed atrial fibrillation with the use of ICM in patients with MINOCA.

To allow for an all-comers data collection, patients with contraindication(s) to ICM implantation will be enrolled into the non-ICM group to assess the frequency of underlying causes of MINOCA and clinical outcomes throughout 5 years.

ELIGIBILITY:
Inclusion Criteria ICM group

1. ≥18 years of age
2. Written informed consent
3. Acute myocardial infarction (AMI) type 1 in accordance with the 4th universal definition of myocardial infarction
4. Non-obstructive coronary arteries on angiography defined as the absence of coronary artery stenoses ≥50% in any potential infarct-related artery
5. No clinically overt specific cause for the acute presentation
6. Subendocardial or transmural late gadolinum enhancement (LGE) consistent with an ischemic etiology on cardiac magnetic resonance imaging (CMR)
7. No clear underlying cause of MINOCA and therefore increased probability of atrial fibrillation

Exclusion Criteria ICM group:

1. Known atrial fibrillation or atrial flutter
2. History of atrial fibrillation or atrial flutter ablation
3. Known coronary artery disease
4. Previous MI
5. Previous percutaneous coronary intervention (PCI)
6. Previous coronary artery bypass grafting (CABG)
7. Contraindications to CMR (i.e. non-MR-compatible implantable cardiac device, glomerular filtration rate (GFR) <30 ml/min)
8. Contraindications to ICM implantation
9. Clear underlying cause of MINOCA before ICM implantation

Inclusion Criteria non-ICM group:

1. ≥18 years of age
2. Written informed consent
3. AMI type 1 in accordance with the 4th universal definition of myocardial infarction
4. Non-obstructive coronary arteries on angiography defined as the absence of coronary artery stenoses ≥50% in any potential infarct-related artery
5. No clinically overt specific cause for the acute presentation
6. Subendocardial or transmural LGE consistent with an ischemic etiology on CMR

Exclusion Criteria non-ICM group:

1. Known coronary artery disease
2. Previous MI
3. Previous PCI
4. Previous CABG
5. Contraindications to CMR (i.e. non-MR-compatible implantable cardiac device, GFR <30 ml/min)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with cardiac magnetic resonance imaging (CMR) confirmed MINOCA at 2 large tertiary care centers in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2031-05-15 (Estimated)

PRIMARY OUTCOMES:
ICM group: Atrial fibrillation | 1 year
  The occurrence of first diagnosed atrial fibrillation in patients with MINOCA according to ICM
Non-ICM group: Frequency of underlying causes of MINOCA | 1 year
  The frequency of underlying causes of MINOCA (i.e. plaque rupture, plaque erosion, coronary thrombus, coronary dissection, eruptive calcific nodule, coronary spasm (including microvascular dysfunction), coronary thromboembolism due to intra- or extracardiac sources of thrombi (including thromboembolism in the context of a persistent foramen ovale (PFO)), atrial fibrillation according to 3 7-day-Holter-ECGs, other sources of coronary embolism (e.g. vegetations, complex aortic plaques), and arterial thrombophilia

SECONDARY OUTCOMES:
ICM group: Time to first diagnosed atrial fibrillation | ~2 years (battery end of life or explantation of ICM)
  Time to first occurrence of atrial fibrillation according to ICM
ICM group: Time to different durations of first diagnosed atrial fibrillation | ~2 years (battery end of life or explantation of ICM)
  Time to first diagnosis of atrial fibrillation (lasting ≥30 seconds; ≥6 minutes; ≥1 hour; ≥ 24 hour)
ICM group: Atrial fibrillation burden | ~2 years (battery end of life or explantation of ICM)
  Time spent in atrial fibrillation divided by total rhythm monitoring time x100 (%)
ICM group: First diagnosis of atrial fibrillation, stroke or death | 1 year
  Time to composite of first diagnosis of atrial fibrillation, stroke or death
ICM group: Other brady- or tachyarrhythmias | ~2 years (battery end of life or explantation of ICM)
  The incidence and time to first occurrence of other brady- or tachyarrhythmias
ICM group: Predictive value of CMR parameters for atrial fibrillation | ~2 years (battery end of life or explantation of ICM)
  Predictive value of atrial parameters of CMR imaging for the diagnosis of atrial fibrillation
ICM group: Frequency of non atrial fibrillation related etiologies of MINOCA | 1 year
  The frequency of non atrial fibrillation related etiologies of MINOCA (i.e. plaque rupture, plaque erosion, coronary thrombus, coronary dissection, eruptive calcific nodule, coronary spasm (including microvascular dysfunction), coronary thromboembolism due to other intra- or extracardiac sources of thrombi not related to atrial fibrillation (including thromboembolism in the context PFO), other sources of coronary embolism (e.g. vegetations, complex aortic plaques), and arterial thrombophilia
Both groups: Clinical outcomes | 5 years
  The occurrence of all-cause death, cardiac death, myocardial infarction, coronary revascularization, stroke, transitory ischemic attack, deep vein thrombosis, pulmonary embolism, and systemic arterial thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, MD, PhD, Principal Investigator — Bern University Hospital Inselspital
Locations (2):
- Switzerland (2):
  - Bern University Hospital Inselspital, Bern
  - University Hospital Zurich USZ, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agewall S, Beltrame JF, Reynolds HR, Niessner A, Rosano G, Caforio AL, De Caterina R, Zimarino M, Roffi M, Kjeldsen K, Atar D, Kaski JC, Sechtem U, Tornvall P; WG on Cardiovascular Pharmacotherapy. ESC working group position paper on myocardial infarction with non-obstructive coronary arteries. Eur Heart J. 2017 Jan 14;38(3):143-153. doi: 10.1093/eurheartj/ehw149. No abstract available. PMID 28158518
- [Background] Tamis-Holland JE, Jneid H, Reynolds HR, Agewall S, Brilakis ES, Brown TM, Lerman A, Cushman M, Kumbhani DJ, Arslanian-Engoren C, Bolger AF, Beltrame JF; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; and Council on Quality of Care and Outcomes Research. Contemporary Diagnosis and Management of Patients With Myocardial Infarction in the Absence of Obstructive Coronary Artery Disease: A Scientific Statement From the American Heart Association. Circulation. 2019 Apr 30;139(18):e891-e908. doi: 10.1161/CIR.0000000000000670. PMID 30913893
- [Background] Diederichsen SZ, Haugan KJ, Kronborg C, Graff C, Hojberg S, Kober L, Krieger D, Holst AG, Nielsen JB, Brandes A, Svendsen JH. Comprehensive Evaluation of Rhythm Monitoring Strategies in Screening for Atrial Fibrillation: Insights From Patients at Risk Monitored Long Term With an Implantable Loop Recorder. Circulation. 2020 May 12;141(19):1510-1522. doi: 10.1161/CIRCULATIONAHA.119.044407. Epub 2020 Mar 2. PMID 32114796
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Smilowitz NR, Mahajan AM, Roe MT, Hellkamp AS, Chiswell K, Gulati M, Reynolds HR. Mortality of Myocardial Infarction by Sex, Age, and Obstructive Coronary Artery Disease Status in the ACTION Registry-GWTG (Acute Coronary Treatment and Intervention Outcomes Network Registry-Get With the Guidelines). Circ Cardiovasc Qual Outcomes. 2017 Dec;10(12):e003443. doi: 10.1161/CIRCOUTCOMES.116.003443. PMID 29246884
- [Background] Pasupathy S, Air T, Dreyer RP, Tavella R, Beltrame JF. Systematic review of patients presenting with suspected myocardial infarction and nonobstructive coronary arteries. Circulation. 2015 Mar 10;131(10):861-70. doi: 10.1161/CIRCULATIONAHA.114.011201. Epub 2015 Jan 13. PMID 25587100
- [Background] Barr PR, Harrison W, Smyth D, Flynn C, Lee M, Kerr AJ. Myocardial Infarction Without Obstructive Coronary Artery Disease is Not a Benign Condition (ANZACS-QI 10). Heart Lung Circ. 2018 Feb;27(2):165-174. doi: 10.1016/j.hlc.2017.02.023. Epub 2017 Mar 30. PMID 28408093
- [Background] Safdar B, Spatz ES, Dreyer RP, Beltrame JF, Lichtman JH, Spertus JA, Reynolds HR, Geda M, Bueno H, Dziura JD, Krumholz HM, D'Onofrio G. Presentation, Clinical Profile, and Prognosis of Young Patients With Myocardial Infarction With Nonobstructive Coronary Arteries (MINOCA): Results From the VIRGO Study. J Am Heart Assoc. 2018 Jun 28;7(13):e009174. doi: 10.1161/JAHA.118.009174. PMID 29954744
- [Background] Montenegro Sa F, Ruivo C, Santos LG, Antunes A, Saraiva F, Soares F, Morais J. Myocardial infarction with nonobstructive coronary arteries: a single-center retrospective study. Coron Artery Dis. 2018 Sep;29(6):511-515. doi: 10.1097/MCA.0000000000000619. PMID 29608443
- [Background] Abdu FA, Liu L, Mohammed AQ, Luo Y, Xu S, Auckle R, Xu Y, Che W. Myocardial infarction with non-obstructive coronary arteries (MINOCA) in Chinese patients: Clinical features, treatment and 1 year follow-up. Int J Cardiol. 2019 Jul 15;287:27-31. doi: 10.1016/j.ijcard.2019.02.036. Epub 2019 Feb 20. PMID 30826195
- [Background] Reynolds HR, Maehara A, Kwong RY, Sedlak T, Saw J, Smilowitz NR, Mahmud E, Wei J, Marzo K, Matsumura M, Seno A, Hausvater A, Giesler C, Jhalani N, Toma C, Har B, Thomas D, Mehta LS, Trost J, Mehta PK, Ahmed B, Bainey KR, Xia Y, Shah B, Attubato M, Bangalore S, Razzouk L, Ali ZA, Merz NB, Park K, Hada E, Zhong H, Hochman JS. Coronary Optical Coherence Tomography and Cardiac Magnetic Resonance Imaging to Determine Underlying Causes of Myocardial Infarction With Nonobstructive Coronary Arteries in Women. Circulation. 2021 Feb 16;143(7):624-640. doi: 10.1161/CIRCULATIONAHA.120.052008. Epub 2020 Nov 14. PMID 33191769